CLINICAL TRIAL: NCT02514135
Title: Intra-abdominal Hypertension in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Patrick Murphy, Resident, Western University, Canada
Other Study IDs: WesternUCanada
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Intra-Abdominal Hypertension; Abdominal Compartment Syndrome
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Elevated Intra-abdominal Pressure: Patients with intra-abdominal pressure > 12 mmHg at any time throughout admission
  Interventions: Other: No intervention
- Normal Intra-abdominal Pressure: Patients with intra-abdominal pressure < 12 mmHg throughout admission
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The aim of the proposed study is to determine the incidence and prevalence of intra-abdominal hypertension and abdominal compartment syndrome in consecutive intensive care admissions using broad inclusion criteria.

DETAILED DESCRIPTION:
Increased pressure within the abdominal cavity is particularly common in intensive care patients and has been shown to be an independent risk-factor for mortality in this patient population. The quoted rates of intra-abdominal hypertension of range anywhere from 20-60% are dependent on the population of patient studied. The prospective observational studies performed to date have been underpowered, used strict inclusion/exclusion criteria or were performed prior to consensus guidelines on the definition and measurement of intra-abdominal pressure and hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Foley catheter in-situ on admission

Exclusion Criteria:

* Contra-indication to bladder pressure measurement
* Home service asked that patient is not included
* Death within 24 priors of admission before bladder pressure measured
* No bladder pressure performed within 24 hours of admission
* Consent refused or unable to be obtained (lack of SDM, patient unable to provide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults (>18 years of age) admitted to the intensive care unit at Victoria Hospital, London, Ontario who have a Foley catheter in-situ
Sampling Method: Non-Probability Sample
Enrollment: 286 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-01-30 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Mortality | While patient in-hospital, expected stay one week on average
  As measured prospectively by patient death in the ICU

SECONDARY OUTCOMES:
Length of stay | While patient in-hospital, expected stay one week on average
  Measured prospectively from date of admission to ICU to death, or discharge from ICU
Abdominal decompression | While patient in-hospital, expected stay one week on average
  Midline laparotomy for abdominal compartment syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Kelly N Vogt, MD, Principal Investigator — Western University
Locations (1):
- Victoria Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Kirkpatrick AW, Roberts DJ, De Waele J, Jaeschke R, Malbrain ML, De Keulenaer B, Duchesne J, Bjorck M, Leppaniemi A, Ejike JC, Sugrue M, Cheatham M, Ivatury R, Ball CG, Reintam Blaser A, Regli A, Balogh ZJ, D'Amours S, Debergh D, Kaplan M, Kimball E, Olvera C; Pediatric Guidelines Sub-Committee for the World Society of the Abdominal Compartment Syndrome. Intra-abdominal hypertension and the abdominal compartment syndrome: updated consensus definitions and clinical practice guidelines from the World Society of the Abdominal Compartment Syndrome. Intensive Care Med. 2013 Jul;39(7):1190-206. doi: 10.1007/s00134-013-2906-z. Epub 2013 May 15. PMID 23673399